CLINICAL TRIAL: NCT05099549
Title: A Phase 1/2a, Open-Label, Multi-Center Study Evaluating the Safety, Tolerability, and Anti-Tumor Activity of AFM24 in Combination With Ex Vivo Expanded Autologous Natural Killer Cells (SNK01) in Subjects With Advanced/Metastatic EGFR-Expressing Cancers
Brief Title: Safety, Tolerability, and Anti-Tumor Activity of AFM24 in Combination With SNK01 in Subjects With Advanced/Metastatic EGFR-Expressing Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Affimed and NKGen have mutually decided to discontinue the study. Affimed will evaluate the best options to advance this project with an allogeneic off-the-shelf NK cell product while NKGen will focus on CNS with SNK01.
Sponsor: NKGen Biotech, Inc. (Industry)
Collaborators: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AFM24-SNK01-103
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Advanced Solid Tumor; Refractory Tumor; Metastatic Tumor
Keywords: EGFR Positive; EGFR; EGFR+; AFM24; SNK01; Solid tumor; Lung cancer; Refractory; Metastatic; NSCLC; SCCHN; NK cells; Natural killer cell; IgG1; antibody; CD16A; ADCC; ADCP
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Neoplasms; Neoplasm Metastasis; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled sequentially in cohorts of 3 to 6 subjects into Phase 1/dose escalation. The dose escalation will follow the standard oncology Phase 1 3 + 3 dose escalation design. A minimum of 3 cohorts will be utilized and dose increases will be determined by the Safety Review Committee.
  Once RP2D is determined in Phase 1/dose escalation, the Phase 2a/expansion phase will begin enrolling up to 121 subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1, Dose Escalation (Experimental): It is estimated that approximately 3-6 subjects will be enrolled per cohort in three dose cohorts for a total of 12-18 participants.
  SNK01 (fixed dose) will be administered weekly by IV infusion.
  Interventions: Drug: AFM24; Biological: SNK01
- Phase 2a, Expansion Cohort 1 - Metastatic colorectal cancer (EXP-1: mCRC) (Experimental): SNK01 (fixed dose) will be administered weekly by IV infusion.
  Interventions: Drug: AFM24; Biological: SNK01
- Phase 2a, Expansion Cohort 2 - Head and Neck Squamous Cell Carcinoma (EXP-2: SCCHN) (Experimental): SNK01 (fixed dose) will be administered weekly by IV infusion.
  Interventions: Drug: AFM24; Biological: SNK01
- Phase 2a, Expansion Cohort 3 - Non-small cell lung cancer (EXP-3: NSCLC) (Experimental): SNK01 (fixed dose) will be administered weekly by IV infusion.
  Interventions: Drug: AFM24; Biological: SNK01

INTERVENTIONS:
Drug: AFM24 — Tetravalent, bispecific EGFR- and CD16A-binding innate cell engager.
Biological: SNK01 — Patient-specific ex-vivo expanded autologous natural killer cells.

SUMMARY:
This is an open-label, multi-center study to evaluate the safety, tolerability, and anti-tumor activity of SNK01 in combination with AFM24 in subjects with advanced or metastatic EGFR-expressing cancers.

DETAILED DESCRIPTION:
The study will be conducted in two phases. The Phase 1/dose escalation phase will gather preliminary safety and tolerability data for escalating doses of AFM24 in combination with SNK01 at a fixed dose in order to determine the MTD/RP2D for the combination dose regimen to be used in the Phase 2a/expansion.

The Phase 2a/expansion portion of the study will gather additional safety, tolerability, efficacy, and anti-tumor activity information for the combination of AFM24 with SNK01 in subjects with three types of advanced or metastatic EGFR-expressing cancers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Capable of giving signed informed consent
2. Males and females age ≥ 18 years
3. Phase 1/Dose Escalation : any histologically confirmed advanced or metastatic EGFR-positive malignancy for which all standard of care treatment options have been received and are no longer effective or are considered inappropriate at the discretion of the investigator.
4. Phase 2a/Expansion : histologically confirmed advanced or metastatic EGFR positive malignancy of mCRC (EXP-1 cohort), SCCHN (EXP-2 cohort) or NSCLC (EXP-3 cohort).
5. Additional Criteria for Phase 2a/Expansion: subjects must have a disease history specific to their disease as listed below:

   1. EXP-1: mCRC. Metastatic colorectal cancer (mCRC) MSI low/DNA mismatch repair proficient. Subjects must have received ≥ 1 lines of previous combination therapy and must have been exposed to oxaliplatin, irinotecan, a fluoropyrimidine, a VEGF targeting agent and, if considered appropriate by the treating physician, an EGFR targeted antibody.
   2. EXP-2: SCCHN. Subjects with advanced or metastatic SCCHN whose disease has progressed after having received ≥ 1 prior lines of therapy for advanced disease, which must have included platinum-based therapy, fluoropyrimidine, and an anti PD 1/PD-L1 antibody.
   3. EXP-3: NSCLC. Subjects with advanced or metastatic EGFR-expressing NSCLC (EGFR WT) whose disease has progressed after having received ≥ 1 prior lines of therapy for advanced disease. Subjects must have received at least a platinum-based doublet in combination with anti-PD1/PD-L1 antibody or must have received a platinum-based doublet followed by an anti-PD1/PD-L1 antibody.
6. One or more measurable tumors lesions per RECIST v1.1
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Adequate bone marrow, hepatic and renal function.

Key Exclusion Criteria:

1. Superior vena cava syndrome contra-indicating hydration
2. Untreated or symptomatic central nervous system (CNS) metastases
3. No resolution of specific toxicities related to any prior anti-cancer therapy to Grade ≤ 1 according to the NCI-CTCAE v.5.0 (except peripheral or motor neuropathy, lymphopenia and alopecia)
4. Treatment with systemic anticancer therapy or an investigational device within 4 weeks (6 weeks if therapy was mitomycin C and/or nitrosoureas), or within 5 half-lives of the agent (if half-life is known and it is shorter) before the first dose of study treatment.
5. Radiation therapy within 2 weeks before first dose of any study treatment or unresolved (NCI CTCAE v5.0 Grade > 1) toxicity from previous radiotherapy
6. Clinically significant cardiovascular disease
7. Major surgery within 4 weeks prior to any study treatment administration
8. Any pulmonary, thyroid, renal, hepatic severe/uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol
9. Active uncontrolled viral, fungal, or bacterial infection requiring systematic therapy within 14 days prior to first dose of study treatment.
10. Known history of testing positive for human immunodeficiency virus (HIV), and/or positive test for Hepatitis B virus surface antigen (HBsAg) and/or positive Hep C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection.
11. Autoimmune disease requiring therapy; immunodeficiency, or any disease process requiring systemic immunosuppressive therapy
12. A serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor
13. Any other condition that, in the opinion of the Investigator, would prohibit the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Determine the maximum tolerated dose (MTD) of AFM24 in combination with SNK01. To be assessed by the incidence and severity of dose-limiting toxicity (DLT) within the DLT observation period.
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Determine the recommended phase 2 dose (RP2D) of AFM24 in combination with SNK01.
  To be assessed by the incidence and severity of dose-limiting toxicity (DLT) within the DLT observation period.
Phase 2a/Expansion | Up to 24 months
  Determine objective response rate (ORR) of AFM24 in combination with SNK01. Determine ORR using Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1

SECONDARY OUTCOMES:
Phase 1/Dose Escalation | Up to 24 months
  Assess safety and tolerability of AFM24 in combination with SNK01. Determine frequency and severity of treatment-emergent AEs (TEAEs) per National Cancer Institute's Common Toxicity Criteria for Adverse Events (NCI CTCAE v 5.0).
Phase 1/Dose Escalation | Up to 24 months
  Determine preliminary efficacy of AFM24 in combination with SNK01. Determine ORR using RECIST v1.1 evaluated by local assessment.
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Maximum observed plasma concentration (Cmax) of AFM24
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Time to maximum plasma concentration (Tmax) of AFM24
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Minimum plasma concentration (Cmin) of AFM24
Phase 1/Dose Escalation | 28 days starting on cycle 1 day 1
  Area under plasma concentration-time curve for dosing interval (AUCtau) of AFM24
Phase 1/Dose Escalation | Up to 24 months
  Immunogenicity of AFM24 when AFM24 is given in combination with SNK01 Frequency of subjects developing AFM24 anti drug antibodies (ADAs) through completion of the Phase 1/dose escalation portion
Phase 2a/Expansion | Up to 24 months
  Safety and tolerability of AFM24 in combination with SNK01 Frequency of TEAEs graded according to NCI CTCAE v 5.0
Phase 2a/Expansion | Up to 24 months
  To assess progression-free survival (PFS) according to RECIST v1.1 by local assessment Assess the number of subjects with PFS defined as duration of time from start of combination treatment to date of progression.
Phase 2a/Expansion | Up to 24 months
  To assess overall survival (OS).
Phase 2a/Expansion | Up to 24 months
  To assess duration of response (DOR) according to RECIST v1.1 by local assessment.
Phase 2a/Expansion | Up to 24 months
  To assess clinical benefit rate (CBR) according to RECIST v1.1 by local assessment.
Phase 2a/Expansion | 28 days starting on cycle 1 day 1
  Maximum observed plasma concentration (Cmax) of AFM24.
Phase 2a/Expansion | 28 days starting on cycle 1 day 1
  Time to maximum plasma concentration (Tmax) of AFM24.
Phase 2a/Expansion | 28 days starting on cycle 1 day 1
  Minimum plasma concentration (Cmin) of AFM24.
Phase 2a/Expansion | 28 days starting on cycle 1 day 1
  Area under plasma concentration-time curve for dosing interval (AUCtau) of AFM24.
Phase 2a/Expansion | Up to 24 months
  Immunogenicity of AFM24 when AFM24 is given in combination with SNK01 Frequency of subjects developing AFM24 ADAs and frequency of subjects developing neutralizing ADAs.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chang, MPH, Study Director — NKGen Biotech, Inc.
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Chicago, Chicago, Illinois